CLINICAL TRIAL: NCT07200297
Title: Comparison of Three Different Oral Care Methods in Terms of Oral Health in Intensive Care Patients Receiving Non-Invasive Mechanical Ventilation: A Randomized Controlled Trial
Brief Title: A Comparative Study of Three Oral Care Methods in NIMV Patients in Intensive Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SÜMEYYE BİLGİLİ TEKİN (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, SÜMEYYE BİLGİLİ TEKİN, Nursing Fundamentals Graduate Student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AU-SBİLGİLİ_003
Record Dates: First submitted 2025-09-10; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Oral Complication
Keywords: Toothbrushing; Intensive Care Units; Non-invasive Ventilation; Oral care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator)
  Interventions: Other: Active Comparator: Control
- Electric Toothbrush (Experimental)
  Interventions: Other: Experimental: Electric Toothbrush
- Manual Toothbrush (Experimental)
  Interventions: Other: Experimental: Manual Toothbrush

INTERVENTIONS:
Other: Active Comparator: Control — Patients who were given only a standard chlorhexidine oral care set
  Arms: Control
Other: Experimental: Electric Toothbrush — Patients who were given an electric toothbrush and toothpaste along with a chlorhexidine set
  Arms: Electric Toothbrush
Other: Experimental: Manual Toothbrush — Patients who were given a manual toothbrush and toothpaste along with a chlorhexidine set.
  Arms: Manual Toothbrush

SUMMARY:
This study aims to examine the effects of different oral care methods on oral health in patients receiving non-invasive mechanical ventilation (NIMV) in the intensive care unit. A randomized controlled experimental design will be employed, with three groups: Control Group - patients receiving only the standard chlorhexidine oral care kit; Electric Toothbrush Group - patients receiving the chlorhexidine kit in combination with an electric toothbrush and toothpaste; and Manual Toothbrush Group - patients receiving the chlorhexidine kit along with a manual toothbrush and toothpaste. Data collection tools will include the Patient Demographic Information Form, Oral Assessment Guide, saliva pH measurement, and salivation assessment using the Schirmer Tear Test Strip. The study is designed to compare the effects of different oral care methods on the oral health of patients receiving NIMV and to identify the most effective method.

ELIGIBILITY:
Inclusion Criteria:

* Must be in an intensive care unit
* Must have consented to participate in the study from themselves or their family
* Must be over 18 years of age
* Must be on a non-invasive mechanical ventilator
* Must have no known active infection.
* Must be in a stable state of consciousness and able to communicate.
* Must be expected to remain in intensive care for at least 48 hours.

Exclusion Criteria:

* Intubated patients.
* Patients with severe oral infections or bleeding mucosal wounds.
* Those receiving radiotherapy/chemotherapy to the head and neck region.
* Organ transplant patients.
* Patients without oral anatomic abnormalities or dentures.
* Those who refused to participate in the study or did not sign the consent form.
* Patients with chronic or acute health conditions that prevent oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Oral Health Status | From day 1 to day 3 (3 consecutive days).
  Oral health will be assessed using the Oral Assessment Guide (OAG). The guide examines eight areas (voice, swallowing, lips, tongue, saliva, mucous membranes, gums, and teeth/dentures). Each item is scored from 1 (healthy) to 3 (severely impaired). The total score ranges from 8-24.
  Scale score (8-24). A low score indicates good oral health, while a high score indicates deterioration in oral health.

SECONDARY OUTCOMES:
Saliva pH Value | From day 1 to day 3 (3 consecutive days).
  Saliva pH Value: During the oral health assessment, pH will be measured with an indicator strip.
  Unit of Measurement: pH units (0-14). Neutral pH (≈7) indicates a healthy oral environment. Saliva Production (Salivation): Salivation will be assessed using the Schirmer Tear Test Strip. The strip's wetted length will be recorded.
  Unit of Measurement: Strip wetted in millimeters (mm). Longer wetted length indicates greater saliva production.

CONTACTS AND LOCATIONS:
Overall Officials: Reva PROF.DR, Principal Investigator — https://avesis.atauni.edu.tr/reva
Locations (1):
- Ataturk University, Erzurum, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No